CLINICAL TRIAL: NCT02713321
Title: Impact of Medicaid Health Home on Patients With Diabetes in New York City
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); New York City Clinical Data Research Network (Other); Weill Medical College of Cornell University (Other); The New York Academy of Medicine (Other)
Responsible Party: Principal Investigator, Victoria Mayer, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: GCO 15-1545; NEN-1508-32252 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; vulnerable populations; comorbidity; patient-centered outcomes research; Medicaid reform; health disparities
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Specify all types of biospecimens to be retained (e.g., whole blood, serum, white cells, urine, tissue)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health Home patients: The cohort is made up of patients with type 2 diabetes, insured by Medicaid, and eligible for participation in a Medicaid Health Home (either due to HIV infection, serious mental illness, substance abuse, or multiple chronic conditions). One group will include patients who participate in the Health Home program.
- non-Health Home patients: The second group will include patients who do not participate in the Health Home program, but have type 2 diabetes, are insured by Medicaid, and meet eligibility requirements for the Health Homes.

SUMMARY:
Type 2 diabetes is common in the United States; about 1 in 10 people have the disease. Diabetes can cause devastating health events, such as hospitalizations, kidney failure, blindness, amputation, heart attack, stroke, painful nerve damage (neuropathy), and death. There are many barriers for patients with diabetes that get in the way of controlling risk factors, following recommendations, and getting the care they need from the health system to help prevent these complications; this is especially true for those with other health problems too. Those living in poverty and racial/ethnic minorities are more likely to have complications from diabetes, and less likely to get recommended care from health systems. In order to improve care and outcomes for people with complex medical problems, several states have started the Medicaid Health Home (HH) program, including New York State (NYS) in 2012. This program is for people with two or more chronic health conditions, such as diabetes and heart disease, people with HIV, and people with a serious mental health condition. HHs are meant to manage and coordinate care, by helping health care providers, social service agencies, community-based organizations, and health insurance plans work together. Similar programs have been shown, on a smaller scale, to improve some results for patients with diabetes, such as lab tests indicating level of diabetes control. Studies have not yet looked at how a large program like HHs impacts the way healthcare is delivered and impacts the health events that matter most to patients with diabetes. Also, few studies include stakeholders on the research team, even though they stand to benefit the most from such programs, and have the experience needed as patients, clinicians, advocates, and administrators to guide efforts. The investigators have gathered a research team that includes scientific investigators along with a diverse group of partners, including patients, clinicians, and program administrators. The investigators plan to use two data sources that show what happens to individual patients over time: 1) NYS Medicaid insurance data 2) the New York City-Clinical Data Research Network (NYC-CDRN). The NYC-CDRN has identified a group of patients with diabetes from 7 large health systems; it has also developed a system for putting together the same set of information for each patient, and removing any identifying information. The investigator will look at patients who have diabetes and are part of a HH and study what happened to them over time. The investigator will also look at a comparison group of patients who are very similar to the HH patients, but they did not join a HH, and follow them over time. The investigator will then compare these two groups to each other. The investigator will look at the quality of healthcare they received and their health outcomes. The investigator will focus on health outcomes that are meaningful to patients. This study can provide important knowledge about the effects of the HH program on patients with diabetes.

DETAILED DESCRIPTION:
The current PCORI-funded study is evaluating the impact of the NYS Medicaid HH program on the process and outcomes of care for low-income NYC residents with diabetes, compared to non-enrolled residents with similar conditions and utilization histories. The HH program enrolls patients with 1) multiple chronic conditions, 2) serious mental illness, and/or 3) HIV, and provides care management services. The study team now proposes to extend this work to examine the impacts of the pandemic on this vulnerable population, a majority of which is Black or Latinx. The study team hypothesizes that HH participation will reduce pandemic-related disruptions in access to health care and social services and improve health outcomes among patients with diabetes in NYC. Using a quasi-experimental difference-in-differences design, the study team will contrast access and utilization of health care and social services and health outcomes among HH enrollees and non-enrollees during a baseline period prior to the pandemic (CY2019) with each month of the pandemic time period (January- September 2020). In addition, the study team will examine the associations of a range of social determinants and access to health care and social services during the pandemic among low-income patients with clinical diabetes using survey data.

ELIGIBILITY:
Inclusion Criteria:

* adults over age 18
* Type II diabetes
* insured by Medicaid
* low income
* data included in the New York City Clinical Data Research Network (NYC-CDRN)
* for intervention group,Health Home enrollment
* comparison group will be obtained through propensity score matching

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with data in the New York City Clinical Data Research Network (NYC-CDRN). The NYC-CDRN brings together 22 organizations, including 7 independent health systems (Columbia University College of Physicians and Surgeons, Montefiore Medical Center and Albert Einstein College of Medicine, Mount Sinai Health System and the Icahn School of Medicine, New York-Presbyterian Hospital, New York University Langone Medical Center and New York University School of Medicine, Weill Cornell Medical College, and the Clinical Directors Network). This data network includes longitudinal data from both inpatient and outpatient facilities from throughout New York City.
Sampling Method: Non-Probability Sample
Enrollment: 96759 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria L Mayer, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mayer V, Mijanovich T, Deshpande R, et al. (2024). The Impact of Medicaid Health Homes on Patients with Diabetes. Patient-Centered Outcomes Research Institute (PCORI).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with clinical diabetes were identified from the INSIGHT Clinical Research Network electronic health record (EHR) data from 6 large academic NYC healthcare systems from 2010-2017.
Groups:
- Health Home Patients: The cohort is made up of patients with type 2 diabetes, insured by Medicaid, and eligible for participation in a Medicaid Health Home (either due to HIV infection, serious mental illness, or multiple chronic conditions). This group included patients who participated in the Health Home program.
- Non-Health Home Patients: This group included patients who did participate in the Health Home program, but had type 2 diabetes, were insured by Medicaid, and met eligibility requirements for the Health Homes.
Period: Before Matching/Weighting
Arm/Group | Health Home Patients | Non-Health Home Patients
Started | 11969 | 84790
Completed | 11646 | 73973
Not Completed | 323 | 10817
Period: After Matching/Weighting ****
Arm/Group | Health Home Patients | Non-Health Home Patients
Started | 11646 | 73973
Completed | 11646 | 26601
Not Completed | 0 | 47372

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Health Home Patients | Non-Health Home Patients | Total
Number analyzed (Participants) | 11646 | 26601 | 38247
Age, Customized [Count of Participants; unit: Participants]
  15-44 years | 1986 | 4535 | 6521
  45-64 years | 7287 | 16644 | 23931
  65+ years | 2383 | 5443 | 7826
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6999 | 15987 | 22986
  Male | 4647 | 10614 | 15261
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 5674 | 12960 | 18634
  Non-Hispanic Black | 3488 | 7967 | 11455
  Non-Hispanic White | 1228 | 2804 | 4032
  Other/unknown | 1266 | 2892 | 4158
Medicare [Count of Participants; unit: Participants] | 3841 | 8773 | 12614
SSI due to disability [Count of Participants; unit: Participants] | 5720 | 13066 | 18786
SSI due to age [Count of Participants; unit: Participants] | 2344 | 5355 | 7699
Serious mental illness diagnosis [Count of Participants; unit: Participants] | 6254 | 14285 | 20539
Alcohol or substance use disorder diagnosis [Count of Participants; unit: Participants] | 3136 | 7164 | 10300
Cancer diagnosis [Count of Participants; unit: Participants] | 1831 | 4182 | 6013
HIV diagnosis [Count of Participants; unit: Participants] | 3699 | 8448 | 12147
Number of chronic condition indicator (CCI) [Mean (Standard Deviation); unit: indicators] | 17.0 (9.4) | 17.0 (9.4) | 17.0 (9.4)
Hospitalizations [Mean (Standard Deviation); unit: hospitalizations] | 1.0 (2.1) | 1.0 (2.1) | 1.0 (2.1)
ED visits [Mean (Standard Deviation); unit: visits] | 1.1 (4.0) | 1.1 (4.0) | 1.1 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Enrollees With Diabetes-related Preventable Hospitalizations
Description: Proportion of hospitalizations related to diabetes that could have been prevented. Diabetes-related potentially preventable hospitalizations are admissions to a hospital for certain acute illnesses or worsening chronic conditions that might not have required hospitalization had these conditions been managed successfully by primary care providers in outpatient settings.
Time Frame: Baseline and 12 months
Population: Results for HH enrollees and a matched comparison group of HH non-enrollees
Measure: Count of Participants; unit: Participants
Arm/Group | Health Home Patients | Non-Health Home Patients
Number analyzed (Participants) | 11646 | 26601
Participants
  Baseline | 48 | 109
  12 months | 48 | 90

2. Secondary Outcome: Number of Primary Care Visits
Description: Number of primary care visits to assess the impact of Health Home (HH) enrollment compared to usual care among Medicaid-insured patients with diabetes and other chronic conditions on access to health care and social services and COVID-19 and non-COVID-19 clinical outcomes.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Health Home Patients | Non-Health Home Patients
Number analyzed (Participants) | 11646 | 26601
visits | 10.9 (10.9) | 8.7 (10.9)

3. Secondary Outcome: Number of Months of Medicaid Coverage
Description: Number of months of Medicaid coverage to assess the impact of Health Home (HH) enrollment compared to usual care among Medicaid-insured patients with diabetes and other chronic conditions on access to health care and social services and COVID-19 and non-COVID-19 clinical outcomes.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: months
Groups:
- Health Home Patients: The cohort is made up of patients with type 2 diabetes, insured by Medicaid, and eligible for participation in a Medicaid Health Home (either due to HIV infection, serious mental illness, , or multiple chronic conditions). This group included patients who participated in the Health Home program.
- Non-Health Home Patients: This group included patients who did not participate in the Health Home program, but had type 2 diabetes, were insured by Medicaid, and met eligibility requirements for the Health Homes.
Arm/Group | Health Home Patients | Non-Health Home Patients
Number analyzed (Participants) | 11646 | 26601
months | 11.7 (1.3) | 10.7 (1.3)

ADVERSE EVENTS:
Time Frame: Adverse events not collected
Description: Adverse Events not collected
Arm/Group | Health Home Patients | Non-Health Home Patients
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/21/NCT02713321/Prot_000.pdf